CLINICAL TRIAL: NCT03359850
Title: An Open-Label, Non-Randomized, Multicenter Study to Determine the Pharmacokinetics and Safety of Niraparib Following a Single Oral Dose in Patients With Advanced Solid Tumors and Either Normal Hepatic Function or Moderate Hepatic Impairment
Brief Title: Pharmacokinetic and Safety Study of Niraparib With Normal or Moderate Hepatic Impairment Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 213354; 3000-01-003 (Other: Tesaro)
Record Dates: First submitted 2017-10-03; First posted 2017-12-02 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Ovarian Neoplasms; Neoplasms; Solid Tumor; Hepatic Impairment
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — niraparib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal hepatic function (Group 1): (Experimental): To evaluate the pharmocokinetics and safety of niraparib
  Interventions: Drug: Niraparib
- Moderate hepatic impairment (Group 2): (Experimental): To evaluate the pharmocokinetics and safety of niraparib
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib is a potent, orally active PARP1 and PARP2 inhibitor being developed as a treatment for patients with tumors that harbor defects in the homologous recombination DNA repair pathway or that are driven by PARP-mediated transcription factors.
  Other Names: Zejula®

SUMMARY:
Niraparib (Zejula®)is extensively metabolized and eliminated primarily by hepatic and renal pathways. The purpose of this study is to evaluate pharmacokinetics and safety of niraparib in patients with moderate hepatic impairment, for the purpose of providing recommendations to guide the initial dose and dose titration in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis and Criteria for Inclusion:

All patients:

To be considered eligible to participate in this study, all of the following requirements must be met:

1. Patient, male or female, is at least 18 years of age.
2. Patient has a diagnosis of advanced solid malignancy that has failed standard therapy or for which standard therapy is not likely to provide meaningful benefit, or patient has refused standard therapy.
3. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Patient is able to take oral medications.
5. Female patient, if of childbearing potential, has a negative serum pregnancy test within 72 hours prior to taking study drug and agrees to abstain from activities that could result in pregnancy from enrollment through 120 days after the last dose of study treatment, or be of non-childbearing potential. Non-childbearing potential is defined as (by other than medical reasons):

   * ≥45 years of age and has not had menses for > 1 year.
   * Amenorrheic for < 2 years without a hysterectomy Post hysterectomy, bilateral oophorectomy, or tubal ligation..

   Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
6. Male patient agrees to use an adequate method of contraception starting with the first dose of study treatment through 120 days after the last dose of study treatment..
7. Patient is able to understand the study procedures and agrees to participate in the study by providing written informed consent.

Patients with normal hepatic function (Group 1):

Patients screened for the normal hepatic function group must meet the following additional criteria to be eligible for enrollment:

1. Patient has no history of hepatic impairment.
2. Patient has liver function test (LFT) results within normal range:

   * Total bilirubin ≤ ULN
   * Aspartate aminotransferase (AST) ≤ ULN.
   * INR ≤1.5 X ULN unless the patient is receiving anticoagulant therapy and the INR is within therapeutic range of intended use of anticoagulants.
3. Patient has adequate hematologic and renal function as defined below:

   * Absolute neutrophil count ≥1500/µL
   * Platelets ≥100,000/µL
   * Hemoglobin ≥9 g/dL
   * Serum creatinine ≤1.5 × ULN or a calculated creatinine clearance ≥60 mL/min using the Cockcroft-Gault equation.

Patients with moderate hepatic impairment (Group 2):

Patients screened for the moderate hepatic impairment group must meet the following additional criteria to be eligible for enrollment:

1. Patient has stable, moderate hepatic impairment, defined as:

   * BILI: >1.5 × to 3 × ULN, for at least 2 weeks prior to Day 1
   * AST: Any value
   * INR less than 1.8 unless the patient is receiving anticoagulant therapy and the INR is within therapeutic range of intended use of anticoagulants.
2. Patient has hematologic and renal function as defined below:

   * Absolute neutrophil count ≥1000/µL
   * Platelets ≥75,000/µL
   * Hemoglobin ≥8 g/dL
   * Serum creatinine ≤1.5 × ULN or a calculated creatinine clearance ≥60 mL/min using the Cockcroft-Gault equation.
3. Patient's hepatic disease is deemed stable by the Investigator

Criteria for Exclusion:

Patients will not be eligible for study entry if any of the following criteria are met:

All patients:

1. Patient has undergone palliative radiotherapy within 1 week of study drug administration, encompassing >20% of the bone marrow.
2. Patient is starting chemotherapy within 3 weeks of study drug administration.
3. Patient has a known hypersensitivity to the components of niraparib or excipients
4. Patients who received colony-stimulating factors within 2 weeks prior to the first dose of study treatment are not eligible.
5. Patient has persistent chemotherapy associated Grade 2 or greater toxicity except for neuropathy, alopecia or fatigue.
6. Patient has symptomatic uncontrolled brain or leptomeningeal metastases.
7. Patient has undergone major surgery within 3 weeks of starting the study or patient has not recovered from any effects of any major surgery.
8. Patient is considered a poor medical risk due to a serious, uncontrolled medical disorder (other than hepatic impairment) or active, uncontrolled infection.
9. Patient has received a transfusion (platelets or red blood cells) within 3 weeks of receiving niraparib.
10. Patient is pregnant, breastfeeding, or expecting to conceive children while receiving study treatment or for 3 months after the last dose of study treatment.
11. Patient has a known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

    NOTE: Exclusion Criteria 12-16 apply patients participating in the PK phase of the study.
12. Patient is currently receiving, or unable to refrain from taking from 4 days prior to dosing until the time of the last PK blood draw, any of the following cytochrome (CYP) 1A2 substrates: alosetron, duloxetine, melatonin, ramelteon, tacrine, tizanidine, and theophylline.
13. Patient is unable to refrain from any intake of grapefruit or grapefruit juice within 4 days of the first administration of niraparib until the final PK sample collection.
14. Patient is currently receiving, or unable to refrain from taking from 4 days prior to dosing until the last PK blood draw, any of the following P-glycoprotein (P-gp) inhibitors: amiodarone, azithromycin, captopril, carvedilol, clarithromycin, conivaptan, cyclosporine, diltiazem, dronedarone, erythromycin, felodipine, itraconazole, ketoconazole, lopinavir and ritonavir, quercetin, quinidine, ranolazine, ticagrelor and verapamil.
15. Patient is taking proton pump inhibitors, antacids, or histamine 2 (H2) blockers within 48 hours prior to niraparib administration, and/or within 6 hours after niraparib administration.
16. Patient has esophagogastrointestinal disease or resection that is likely to interfere with the absorption of niraparib.

Patients with moderate hepatic impairment (Group 2):

Patients screened for the moderate hepatic impairment group who meet any of the following additional criteria will be excluded from the study:

1. Patient has hepatic encephalopathy, severe portal hypertension and/or porto-systemic shunt.
2. Patient has fluctuating or rapidly deteriorating hepatic function as determined by the investigator within the screening period.
3. Patient has acute liver disease caused by drug toxicity or by an infection.
4. Patient has biliary obstruction or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
5. Patient has esophageal variceal bleeding within the past 2 months.
6. Patient is receiving anticoagulant therapy with warfarin or related coumarins.
7. Patient has a history of hepatic transplant, systemic lupus erythematosus, or hepatic coma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2020-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akce M, El-Khoueiry A, Piha-Paul SA, Bacque E, Pan P, Zhang ZY, Ewesuedo R, Gupta D, Tang Y, Milton A, Zajic S, Judson PL, O'Bryant CL. Pharmacokinetics and safety of niraparib in patients with moderate hepatic impairment. Cancer Chemother Pharmacol. 2021 Nov;88(5):825-836. doi: 10.1007/s00280-021-04329-8. Epub 2021 Jul 29. PMID 34324028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated pharmacokinetics and safety of niraparib in participants with advanced solid tumors and with either normal hepatic function or moderate hepatic impairment.
Pre-assignment Details: This is a 2 period study including pharmacokinetic (PK) phase and extension (Ext.) phase. A total of 17 participants were enrolled in the study and received study treatment, niraparib.
Groups:
- Participants With Normal Hepatic Function: All participants received a single dose of 300 milligrams (mg) (3X100 mg capsules) niraparib administered on Day 1 of PK phase. Upon entering extension phase, participants with screening actual body weight >= 77 kilograms (kg) and current platelet count of >=150,000 cells per microliter (c/μL) at C1D1 continued to receive niraparib 300 mg/day (3X100 mg) once daily (QD) on Day 1 of every cycle until treatment discontinuation(each cycle of 28-days). Participants with screening actual body weight < 77 kg and/or current platelet count of <150,000 c/μL continued to receive niraparib 200 mg (2X100 mg capsules) QD on Day 1 of every cycle until treatment discontinuation (each cycle of 28 days).
- Participants With Impaired Hepatic Function: All participants received a single dose of 300 mg (3X100 mg capsules) niraparib administered on Day 1 of PK phase. Upon entering extension phase, participants received niraparib 200 mg (2X100 mg capsules) QD on Day 1 of every cycle until treatment discontinuation (each cycle of 28 days).
Period: PK Phase (Up to Day 8)
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Started | 9 | 8
Completed | 8 | 7
Not Completed | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 1 | 0
Period: Extension Phase (Up to 28 Months)
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Started | 8 | 7
Completed | 0 | 1
Not Completed | 8 | 6
Not completed — Death | 2 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Disease Progression | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] — Safety Population consisted of all participants who received drug
  Years | 64.8 (6.69) | 63.6 (7.71) | 64.2 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  White | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Niraparib and Its Major Metabolite (M1) During PK Phase
Description: Blood samples were collected at indicated time points to evaluate AUC (last) of niraparib and M1. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose Day 1
Population: PK population consisted of all participants who have received niraparib and have sufficient evaluable samples
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 8
Hour*nanogram per milliliter (hr*ng/mL)
  Niraparib | 18500 (37.7) | 26800 (49.6)
  M1 | 19000 (27.5) | 12400 (55.0)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC 0-infinity) of Niraparib and M1 During PK Phase
Description: Blood samples were collected at indicated time points to evaluate AUC (0-infinity) of niraparib and M1. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose Day 1
Population: PK population. Only those participants with data available at specified data points were analyzed (represented by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 7
Hour*nanogram per milliliter (hr*ng/mL)
  Niraparib, n= 9, 7 | 19700 (38.7) | 30800 (54.3)
  M1, n=9, 3: number analyzed (Participants) | 9 | 3
  M1, n=9, 3 | 20700 (29.8) | 21500 (25.4)

3. Primary Outcome: Observed Maximum Plasma Concentration (Cmax) of Niraparib and M1 During PK Phase
Description: Blood samples were collected at indicated time points to evaluate Cmax of niraparib and M1. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose Day 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 8
Nanogram per milliliter
  Niraparib | 594 (45.6) | 553 (47.4)
  M1 | 398 (17.6) | 151 (89.3)

4. Primary Outcome: Time to Maximum Concentration (Tmax) of Niraparib and M1 During PK Phase
Description: Blood samples were collected at indicated time points to evaluate tmax of niraparib and M1. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose Day 1
Population: PK population
Measure: Median (Full Range); unit: Hour
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 8
Hour
  Niraparib | 4.00 [3.00 to 6.33] | 4.09 [2.00 to 8.02]
  M1 | 6.00 [4.00 to 12.08] | 17.73 [6.00 to 25.17]

5. Primary Outcome: Terminal Half-life (t½) of Niraparib and M1 During PK Phase
Description: Blood samples were collected at indicated time points to evaluate t1/2 of niraparib and M1. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 7
Hour
  Niraparib, n=9, 7 | 43.9 (11.5) | 54.8 (25.8)
  M1, n=9, 3: number analyzed (Participants) | 9 | 3
  M1, n=9, 3 | 47.9 (16.6) | 43.7 (20.7)

6. Primary Outcome: Apparent Total Body Clearance (CL/F) of Niraparib and M1 During PK Phase
Description: CL/F is calculated as Dose/(AUC 0-inf). Blood samples were collected at indicated time points to evaluate CL/F of niraparib and M1. PK parameters were calculated by standard non-compartmental analysis. Not applicable (NA) indicates that CL/F could not be measured for M1 since the dose of metabolite is unknown and only known dose is that of parent niraparib.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120, 168 hours post dose Day 1
Population: PK population. Only those participants with data available at specified data points were analyzed. CL/F could not be measured for M1 since the dose of metabolite is unknown and only known dose is that of parent niraparib.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 7
Liters per hour
  Niraparib | 15.2 (38.7) | 9.74 (54.3)
  M1 | NA (NA) — NA indicates that CL/F could not be measured for M1 since the dose of metabolite is unknown and only known dose is that of parent niraparib. | NA (NA) — NA indicates that CL/F could not be measured for M1 since the dose of metabolite is unknown and only known dose is that of parent niraparib.

7. Other Pre Specified Outcome: Plasma Protein Unbound Fraction (Fu) of Niraparib and M1 During PK Phase
Description: Unbound fraction is the unbound concentration of niraparib and M1 in plasma divided by total concentration. This analysis was planned but not performed due to insufficient participants with data
Time Frame: Pre-dose, 3 hours and 168 hours post dose Day 1
Population: PK population.
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Clearance of Unbound Niraparib and M1 (CLfu/F) During PK Phase
Description: CLfu/F is the clearance for unbound niraparib and M1. This analysis was planned but not performed due to insufficient participants with data
Time Frame: Pre-dose, 3 hours and 168 hours post dose Day 1
Population: PK population.
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE) Including Non-serious Adverse Events (Non-SAEs), Serious Adverse Events (SAEs) and Discontinuations Due to AEs During PK Phase
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; or is an important medical event(s) requiring medical or scientific judgment. Treatment-emergent are any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment.
Time Frame: Up to Day 8
Population: Safety Population for PK phase consisted of all participants who received atleast one dose of the investigational drug niraparib during the PK phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 8
Participants
  Any Non -SAEs | 5 | 3
  Any SAE | 1 | 0
  Any Discontinuations due to AE | 1 | 0

10. Secondary Outcome: Change From Baseline in Hemoglobin (Hb) During PK Phase
Description: Blood samples were collected from participants for evaluation of Hb. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline and at Day 8
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 8
Grams per liter | -0.5 (7.82) | 0.6 (7.65)

11. Secondary Outcome: Change From Baseline in Platelets, Neutrophils, Monocytes, Lymphocytes and Leukocyte During PK Phase
Description: Blood samples were collected to analyze hematology parameters:Leukocyte, Lymphocytes, Monocytes, Neutrophils and Platelets. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline and Day 8
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 8
10^9 cells per liter
  Lymphocytes | 0.2 (0.38) | -0.1 (0.15)
  Monocytes | 0.1 (0.32) | -0.1 (0.24)
  Neutrophils | -0.5 (2.13) | -0.7 (1.89)
  Platelets | -18.4 (95.41) | -23.4 (60.31)
  Leukocyte | -0.2 (2.04) | -0.8 (2.16)

12. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Protein and Albumin During PK Phase
Description: Blood samples were collected to analyze clinical chemistry parameters: protein and albumin. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline and Day 8
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 8
Grams per liter
  Protein | -1.0 (4.24) | -3.5 (5.55)
  Albumin | -0.9 (2.03) | -2.3 (3.45)

13. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Alkaline Phosphatase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Lactate Dehydrogenase (LDH) During PK Phase
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters: alkaline phosphatase, ALT, AST and LDH. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline and Day 8
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 8
International units per Liter
  Alkaline phosphatase | 26.3 (50.67) | -32.6 (219.03)
  AST | 34.6 (94.42) | -6.4 (43.81)
  ALT | 24.3 (60.82) | -4.4 (10.39)
  LDH | 36.0 (134.66) | -58.5 (137.97)

14. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Amylase During PK Phase
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameter: Amylase. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline and Day 8
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 7
Units per Liter | 74.4 (206.90) | 0.3 (22.92)

15. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Bilirubin and Creatinine During PK Phase
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters: Bilirubin and Creatinine. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline and Day 8
Population: Safety Population. Only those participants with data available at specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 8
Micromoles per liter
  Bilirubin | 0.6 (3.41) | 8.3 (9.47)
  Creatinine | -1.9 (10.87) | -0.7 (17.19)

16. Secondary Outcome: Change From Baseline in Chemistry Parameters: Glucose, Calcium, Chloride, Phosphate, Potassium, Sodium, Magnesium and Blood Urea Nitrogen (BUN) During PK Phase
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameter:Glucose, Calcium, Chloride, Phosphate, Potassium, Sodium, Magnesium and BUN. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline and Day 8
Population: Safety Population. Only those participants with data available at specified data points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 8
Millimoles per liter
  Glucose, n=8, 8 | -0.8 (1.14) | -0.5 (1.61)
  Calcium, n=8, 8 | 0.0 (0.17) | -0.1 (0.15)
  Chloride, n=8, 8 | 1.8 (2.25) | -0.3 (1.83)
  Phosphate, n=8, 8 | 0.1 (0.16) | -0.1 (0.14)
  Potassium, n=8, 8 | -0.2 (0.26) | -0.2 (0.74)
  Sodium, n=8, 8 | 1.6 (2.26) | -0.5 (2.78)
  BUN, n=8, 8 | -0.4 (1.66) | -0.1 (0.97)
  Magnesium, n=8, 7: number analyzed (Participants) | 8 | 7
  Magnesium, n=8, 7 | -0.0 (0.09) | 0.0 (0.09)

17. Secondary Outcome: Change From Baseline in Weight During PK Phase
Description: Weight was measured at indicated time-points. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline, Day 2 and Day 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 8
Kilograms
  Day 2, n=8, 6: number analyzed (Participants) | 8 | 6
  Day 2, n=8, 6 | -0.0 (0.58) | 0.8 (0.87)
  Day 8, n=9, 8 | -0.0 (1.14) | 0.3 (1.30)

18. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) During PK Phase
Description: Vital signs including SBP and DBP were measured at indicated time-points. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline, Day 2 and Day 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 8
Millimeters of mercury
  SBP, Day 2, n=9, 7: number analyzed (Participants) | 9 | 7
  SBP, Day 2, n=9, 7 | 5.9 (10.79) | 5.7 (10.23)
  SBP, Day 8, n=9, 8 | 0.9 (18.58) | 0.3 (9.69)
  DBP, Day 2, n=9, 7: number analyzed (Participants) | 9 | 7
  DBP, Day 2, n=9, 7 | 3.6 (8.38) | 2.7 (3.15)
  DBP, Day 8, n=9, 8 | 2.4 (9.08) | -0.1 (11.18)

19. Secondary Outcome: Change From Baseline in Pulse Rate During PK Phase
Description: Vital sign including pulse rate was measured at indicated time-points. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline, Day 2 and Day 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 8
Beats per minute
  Day 2, n=9, 7: number analyzed (Participants) | 9 | 7
  Day 2, n=9, 7 | 8.9 (11.30) | 1.3 (10.58)
  Day 8, n=9, 8 | 2.8 (11.91) | -2.3 (7.85)

20. Secondary Outcome: Change From Baseline in Body Temperature During PK Phase
Description: Vital sign including body temperature was measured at indicated time-points. Baseline is defined as the most recent measurement prior to the first administration of study drug in PK phase. Change from Baseline was calculated as post dose value minus Baseline value.
Time Frame: Baseline, Day 2 and Day 8
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 9 | 8
Degrees Celsius
  Day 2, n=9, 7: number analyzed (Participants) | 9 | 7
  Day 2, n=9, 7 | -0.0 (0.39) | 0.1 (0.24)
  Day 8, n=9, 8 | 0.1 (0.33) | 0.1 (0.47)

21. Secondary Outcome: Number of Participants With TEAE Including Non-SAEs, SAEs and Discontinuations Due to AEs During Extension Phase
Description: as for outcome 9
Time Frame: Up to 28 months
Population: Safety Population for extension phase consisted of all participants who received atleast one dose of the investigational drug niraparib during the extension phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 7
Participants
  Any Non-SAEs | 8 | 7
  Any SAE | 3 | 2
  Any Discontinuations due to AE | 0 | 1

22. Secondary Outcome: Change From Baseline in Hb During Extension Phase
Description: Blood samples were collected from participants for evaluation of Hb. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 1 (Days 8, 15, 21), Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 5
Grams per liter
  Cycle 1 Day 8, n=8, 5 | 4.3 (5.78) | 1.0 (8.89)
  Cycle 1 Day 15, n=8, 4: number analyzed (Participants) | 8 | 4
  Cycle 1 Day 15, n=8, 4 | -0.5 (6.32) | -8.3 (15.73)
  Cycle 1 Day 21, n=7, 4: number analyzed (Participants) | 7 | 4
  Cycle 1 Day 21, n=7, 4 | -2.6 (12.91) | -22.3 (17.19)
  Cycle 2 Day 1, n=6, 2: number analyzed (Participants) | 6 | 2
  Cycle 2 Day 1, n=6, 2 | -8.0 (14.93) | -15.0 (1.41)
  Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Cycle 3 Day 1, n=3, 1 | -16.7 (12.10) | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 4 Day 1, n=3, 0 | -10.7 (11.06) |
  Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 5 Day 1, n=3, 0 | -3.7 (2.08) |
  Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Cycle 6 Day1, n=2, 0 | 3.0 (7.07) |

23. Secondary Outcome: Change From Baseline in Platelets, Neutrophils, Monocytes, Lymphocytes and Leukocytes During Extension Phase
Description: Blood samples were collected to analyze hematology parameters: Lymphocytes, Leukocytes, Monocytes, Neutrophils and Platelets. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: as for outcome 22
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 8 | 5
10^9 cells per liter
  Lymphocytes, Cycle 1 Day 8, n=7, 5: number analyzed (Participants) | 7 | 5
  Lymphocytes, Cycle 1 Day 8, n=7, 5 | -0.2 (0.36) | -0.1 (0.22)
  Lymphocytes, Cycle 1 Day 15, n=8, 4: number analyzed (Participants) | 8 | 4
  Lymphocytes, Cycle 1 Day 15, n=8, 4 | -0.1 (0.37) | -0.0 (0.48)
  Lymphocytes, Cycle 1 Day 21, n=7, 4: number analyzed (Participants) | 7 | 4
  Lymphocytes, Cycle 1 Day 21, n=7, 4 | -0.1 (0.25) | -0.2 (0.20)
  Lymphocytes, Cycle 2 Day 1, n=6, 2: number analyzed (Participants) | 6 | 2
  Lymphocytes, Cycle 2 Day 1, n=6, 2 | -0.1 (0.33) | 0.1 (0.04)
  Lymphocytes, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Lymphocytes, Cycle 3 Day 1, n=3, 1 | -0.3 (0.24) | 0.2 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Lymphocytes, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Lymphocytes, Cycle 4 Day 1, n=3, 0 | 0.0 (0.33) |
  Lymphocytes, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Lymphocytes, Cycle 5 Day 1, n=3, 0 | 0.3 (0.30) |
  Lymphocytes, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Lymphocytes, Cycle 6 Day1, n=2, 0 | -0.0 (0.54) |
  Monocytes, Cycle 1 Day 8, n=7, 5: number analyzed (Participants) | 7 | 5
  Monocytes, Cycle 1 Day 8, n=7, 5 | -0.1 (0.20) | 0.0 (0.11)
  Monocytes, Cycle 1 Day 15, n=8, 4: number analyzed (Participants) | 8 | 4
  Monocytes, Cycle 1 Day 15, n=8, 4 | -0.2 (0.28) | -0.1 (0.22)
  Monocytes, Cycle 1 Day 21, n=7, 4: number analyzed (Participants) | 7 | 4
  Monocytes, Cycle 1 Day 21, n=7, 4 | -0.2 (0.20) | -0.1 (0.40)
  Monocytes, Cycle 2 Day 1, n=6, 2: number analyzed (Participants) | 6 | 2
  Monocytes, Cycle 2 Day 1, n=6, 2 | -0.1 (0.14) | -0.1 (0.16)
  Monocytes, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Monocytes, Cycle 3 Day 1, n=3, 1 | -0.2 (0.06) | 0.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed
  Monocytes, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Monocytes, Cycle 4 Day 1, n=3, 0 | -0.0 (0.09) |
  Monocytes, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Monocytes, Cycle 5 Day 1, n=3, 0 | -0.1 (0.10) |
  Monocytes, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Monocytes, Cycle 6 Day1, n=2, 0 | -0.1 (0.16) |
  Neutrophils, Cycle 1 Day 8, n=7, 5: number analyzed (Participants) | 7 | 5
  Neutrophils, Cycle 1 Day 8, n=7, 5 | 0.4 (0.87) | 0.4 (0.44)
  Neutrophils, Cycle 1 Day 15, n=8, 4: number analyzed (Participants) | 8 | 4
  Neutrophils, Cycle 1 Day 15, n=8, 4 | 0.3 (1.01) | 0.5 (0.73)
  Neutrophils, Cycle 1 Day 21, n=7, 4: number analyzed (Participants) | 7 | 4
  Neutrophils, Cycle 1 Day 21, n=7, 4 | -0.6 (1.92) | -0.2 (0.81)
  Neutrophils, Cycle 2 Day 1, n=6, 2: number analyzed (Participants) | 6 | 2
  Neutrophils, Cycle 2 Day 1, n=6, 2 | 0.6 (2.03) | -1.8 (1.94)
  Neutrophils, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Neutrophils, Cycle 3 Day 1, n=3, 1 | -0.0 (1.70) | -0.5 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed
  Neutrophils, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Neutrophils, Cycle 4 Day 1, n=3, 0 | -0.4 (0.51) |
  Neutrophils, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Neutrophils, Cycle 5 Day 1, n=3, 0 | 0.5 (0.27) |
  Neutrophils, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Neutrophils, Cycle 6 Day1, n=2, 0 | -0.1 (0.78) |
  Platelets, Cycle 1 Day 8, n=8, 5 | 12.0 (21.75) | -0.8 (21.32)
  Platelets, Cycle 1 Day 15, n=8, 4: number analyzed (Participants) | 8 | 4
  Platelets, Cycle 1 Day 15, n=8, 4 | -58.1 (118.98) | -8.3 (63.33)
  Platelets, Cycle 1 Day 21, n=7, 4: number analyzed (Participants) | 7 | 4
  Platelets, Cycle 1 Day 21, n=7, 4 | -81.9 (113.91) | -19.3 (57.70)
  Platelets, Cycle 2 Day 1, n=6, 2: number analyzed (Participants) | 6 | 2
  Platelets, Cycle 2 Day 1, n=6, 2 | 55.3 (128.24) | -102.5 (130.81)
  Platelets, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Platelets, Cycle 3 Day 1, n=3, 1 | -46.3 (36.46) | 59.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed
  Platelets, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Platelets, Cycle 4 Day 1, n=3, 0 | 34.0 (43.92) |
  Platelets, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Platelets, Cycle 5 Day 1, n=3, 0 | 45.7 (22.68) |
  Platelets, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Platelets, Cycle 6 Day1, n=2, 0 | 34.0 (42.43) |
  Leukocytes, Cycle 1 Day 8, n=8, 5 | 0.4 (1.76) | 0.3 (0.40)
  Leukocytes, Cycle 1 Day 15, n=8, 4: number analyzed (Participants) | 8 | 4
  Leukocytes, Cycle 1 Day 15, n=8, 4 | -0.1 (1.25) | 0.4 (1.28)
  Leukocytes, Cycle 1 Day 21, n=7, 4: number analyzed (Participants) | 7 | 4
  Leukocytes, Cycle 1 Day 21, n=7, 4 | -1.0 (2.05) | -0.5 (1.36)
  Leukocytes, Cycle 2 Day 1, n=6, 2: number analyzed (Participants) | 6 | 2
  Leukocytes, Cycle 2 Day 1, n=6, 2 | 0.5 (1.96) | -1.9 (1.91)
  Leukocytes, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Leukocytes, Cycle 3 Day 1, n=3, 1 | -0.5 (1.67) | -0.2 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed
  Leukocytes, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Leukocytes, Cycle 4 Day 1, n=3, 0 | -0.4 (0.76) |
  Leukocytes, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Leukocytes, Cycle 5 Day 1, n=3, 0 | 0.9 (0.31) |
  Leukocytes, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Leukocytes, Cycle 6 Day1, n=2, 0 | -0.3 (1.48) |

24. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Protein and Albumin During Extension Phase
Description: Blood samples were collected to analyze clinical chemistry parameters: protein and albumin. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 6 | 2
Grams per liter
  Protein, Cycle 2 Day 1, n=6, 2 | -1.0 (6.96) | -2.0 (0.00)
  Protein, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Protein, Cycle 3 Day 1, n=3, 1 | -2.0 (3.46) | -5.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Protein, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Protein, Cycle 4 Day 1, n=3, 0 | 1.0 (3.61) |
  Protein, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Protein, Cycle 5 Day 1, n=3, 0 | 4.0 (2.65) |
  Protein, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Protein, Cycle 6 Day1, n=2, 0 | 0.0 (2.83) |
  Albumin, Cycle 2 Day 1, n=6, 2 | 0.3 (4.37) | -1.0 (0.00)
  Albumin, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Albumin, Cycle 3 Day 1, n=3, 1 | 1.0 (2.65) | -1.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Albumin, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Albumin, Cycle 4 Day 1, n=3, 0 | 2.7 (3.21) |
  Albumin, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Albumin, Cycle 5 Day 1, n=3, 0 | 4.7 (2.52) |
  Albumin, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Albumin, Cycle 6 Day1, n=2, 0 | 17.0 (16.97) |

25. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Alkaline Phosphatase, ALT, AST and LDH During Extension Phase
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameters: alkaline phosphatase, ALT, AST and LDH. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 6 | 2
International units per Liter
  Alkaline Phosphatase, Cycle 2 Day 1, n=6, 2 | 23.3 (17.43) | -53.5 (221.32)
  Alkaline Phosphatase, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Alkaline Phosphatase, Cycle 3 Day 1, n=3, 1 | 19.7 (5.03) | 57.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Alkaline Phosphatase, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Alkaline Phosphatase, Cycle 4 Day 1, n=3, 0 | 20.0 (10.54) |
  Alkaline Phosphatase, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Alkaline Phosphatase, Cycle 5 Day 1, n=3, 0 | 12.0 (14.80) |
  Alkaline Phosphatase, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Alkaline Phosphatase, Cycle 6 Day1, n=2, 0 | 1.5 (16.26) |
  ALT, Cycle 2 Day 1, n=6, 2 | 11.8 (19.77) | -6.5 (20.51)
  ALT, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  ALT, Cycle 3 Day 1, n=3, 1 | 4.7 (6.11) | 4.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  ALT, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  ALT, Cycle 4 Day 1, n=3, 0 | 2.0 (5.00) |
  ALT, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  ALT, Cycle 5 Day 1, n=3, 0 | 5.3 (7.02) |
  ALT, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  ALT, Cycle 6 Day1, n=2, 0 | 2.0 (4.24) |
  AST, Cycle 2 Day 1, n=6, 2 | 4.8 (5.81) | -25.0 (38.18)
  AST, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  AST, Cycle 3 Day 1, n=3, 1 | 2.0 (2.65) | 4.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  AST, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  AST, Cycle 4 Day 1, n=3, 0 | 4.3 (2.31) |
  AST, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  AST, Cycle 5 Day 1, n=3, 0 | 5.3 (2.52) |
  AST, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  AST, Cycle 6 Day1, n=2, 0 | 5.5 (4.95) |
  LDH, Cycle 2 Day 1, n=3, 2: number analyzed (Participants) | 3 | 2
  LDH, Cycle 2 Day 1, n=3, 2 | 11.7 (37.53) | -625.0 (847.11)
  LDH, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  LDH, Cycle 3 Day 1, n=3, 1 | 6.7 (17.56) | -9.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  LDH, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  LDH, Cycle 4 Day 1, n=3, 0 | -11.7 (41.77) |
  LDH, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  LDH, Cycle 5 Day 1, n=3, 0 | -5.3 (21.46) |
  LDH, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  LDH, Cycle 6 Day1, n=2, 0 | 19.0 (35.36) |

26. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Amylase During Extension Phase
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameter: Amylase. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 4 | 2
Units per Liter
  Cycle 2 Day 1, n=4, 2 | -1.0 (16.39) | -2.5 (6.36)
  Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Cycle 3 Day 1, n=3, 1 | -7.0 (14.18) | -4.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 4 Day 1, n=3, 0 | -2.3 (16.77) |
  Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 5 Day 1, n=3, 0 | 3.0 (5.57) |
  Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Cycle 6 Day1, n=2, 0 | -2.5 (31.82) |

27. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Bilirubin and Creatinine During Extension Phase
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameter: Bilirubin and Creatinine. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 6 | 2
Micromoles per liter
  Bilirubin, Cycle 2 Day 1, n=6, 2 | 0.9 (1.79) | -6.0 (8.46)
  Bilirubin, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Bilirubin, Cycle 3 Day 1, n=3, 1 | 0.6 (2.61) | 1.7 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Bilirubin, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Bilirubin, Cycle 4 Day 1, n=3, 0 | 0.6 (0.99) |
  Bilirubin, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Bilirubin, Cycle 5 Day 1, n=3, 0 | 2.9 (0.99) |
  Bilirubin, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Bilirubin, Cycle 6 Day1, n=2, 0 | -0.9 (1.21) |
  Creatinine, Cycle 2 Day 1, n=6, 2 | 7.5 (17.93) | 18.1 (3.13)
  Creatinine, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Creatinine, Cycle 3 Day 1, n=3, 1 | 13.0 (5.03) | 0.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Creatinine, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Creatinine, Cycle 4 Day 1, n=3, 0 | 0.9 (9.56) |
  Creatinine, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Creatinine, Cycle 5 Day 1, n=3, 0 | 5.6 (2.84) |
  Creatinine, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Creatinine, Cycle 6 Day1, n=2, 0 | 5.7 (5.63) |

28. Secondary Outcome: Change From Baseline in Chemistry Parameters: Glucose, Calcium, Chloride, Phosphate, Potassium, Sodium, Magnesium and BUN During Extension Phase
Description: Blood samples were collected at indicated time-points for analysis of clinical chemistry parameter:Glucose, Calcium, Chloride, Phosphate, Potassium, Sodium, Magnesium and BUN. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 6 | 2
Millimoles per liter
  Glucose, Cycle 2 Day 1, n=6, 2 | -0.0 (1.45) | 1.6 (0.47)
  Glucose, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Glucose, Cycle 3 Day 1, n=3, 1 | 0.7 (1.50) | -2.3 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Glucose, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Glucose, Cycle 4 Day 1, n=3, 0 | -0.4 (0.95) |
  Glucose, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Glucose, Cycle 5 Day 1, n=3, 0 | -0.7 (0.90) |
  Glucose, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Glucose, Cycle 6 Day1, n=2, 0 | -0.8 (0.90) |
  Calcium, Cycle 2 Day 1, n=6, 2 | -0.0 (0.16) | 0.0 (0.14)
  Calcium, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Calcium, Cycle 3 Day 1, n=3, 1 | 0.0 (0.06) | 0.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Calcium, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Calcium, Cycle 4 Day 1, n=3, 0 | 0.0 (0.00) |
  Calcium, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Calcium, Cycle 5 Day 1, n=3, 0 | 0.1 (0.10) |
  Calcium, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Calcium, Cycle 6 Day1, n=2, 0 | -0.0 (0.02) |
  Chloride, Cycle 2 Day 1, n=6, 2 | -1.7 (2.25) | -3.5 (2.12)
  Chloride, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Chloride, Cycle 3 Day 1, n=3, 1 | -2.0 (3.61) | 0.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Chloride, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Chloride, Cycle 4 Day 1, n=3, 0 | -0.7 (1.53) |
  Chloride, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Chloride, Cycle 5 Day 1, n=3, 0 | -1.7 (1.15) |
  Chloride, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Chloride, Cycle 6 Day1, n=2, 0 | -2.5 (2.12) |
  Phosphate, Cycle 2 Day 1, n=5, 2: number analyzed (Participants) | 5 | 2
  Phosphate, Cycle 2 Day 1, n=5, 2 | -0.2 (0.34) | 0.3 (0.02)
  Phosphate, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Phosphate, Cycle 3 Day 1, n=3, 1 | 0.0 (0.18) | -0.1 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Phosphate, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Phosphate, Cycle 4 Day 1, n=3, 0 | -0.1 (0.26) |
  Phosphate, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Phosphate, Cycle 5 Day 1, n=3, 0 | 0.0 (0.43) |
  Phosphate, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Phosphate, Cycle 6 Day1, n=2, 0 | 0.0 (0.30) |
  Potassium, Cycle 2 Day 1, n=6, 2 | -0.2 (0.12) | 0.1 (0.21)
  Potassium, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Potassium, Cycle 3 Day 1, n=3, 1 | 0.1 (0.30) | 0.4 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Potassium, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Potassium, Cycle 4 Day 1, n=3, 0 | 0.0 (0.20) |
  Potassium, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Potassium, Cycle 5 Day 1, n=3, 0 | 0.1 (0.38) |
  Potassium, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Potassium, Cycle 6 Day1, n=2, 0 | 0.1 (0.21) |
  Sodium, Cycle 2 Day 1, n=6, 2 | -1.8 (1.17) | -1.5 (2.12)
  Sodium, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Sodium, Cycle 3 Day 1, n=3, 1 | -3.0 (1.73) | 1.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Sodium, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Sodium, Cycle 4 Day 1, n=3, 0 | -1.0 (1.73) |
  Sodium, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Sodium, Cycle 5 Day 1, n=3, 0 | -1.7 (0.58) |
  Sodium, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Sodium, Cycle 6 Day1, n=2, 0 | -1.5 (2.12) |
  BUN, Cycle 2 Day 1, n=6, 2 | 0.3 (2.15) | 1.8 (0.50)
  BUN, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  BUN, Cycle 3 Day 1, n=3, 1 | 0.7 (2.14) | 1.4 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  BUN, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  BUN, Cycle 4 Day 1, n=3, 0 | -1.0 (0.90) |
  BUN, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  BUN, Cycle 5 Day 1, n=3, 0 | -0.5 (1.25) |
  BUN, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  BUN, Cycle 6 Day1, n=2, 0 | -0.5 (0.76) |
  Magnesium, Cycle 2 Day 1, n=5, 2: number analyzed (Participants) | 5 | 2
  Magnesium, Cycle 2 Day 1, n=5, 2 | -0.0 (0.09) | 0.0 (0.00)
  Magnesium, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Magnesium, Cycle 3 Day 1, n=3, 1 | -0.0 (0.04) | 0.1 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Magnesium, Cycle 4 Day 1, n=2, 0: number analyzed (Participants) | 2 | 0
  Magnesium, Cycle 4 Day 1, n=2, 0 | 0.0 (0.00) |
  Magnesium, Cycle 5 Day 1, n=2, 0: number analyzed (Participants) | 2 | 0
  Magnesium, Cycle 5 Day 1, n=2, 0 | 0.1 (0.00) |
  Magnesium, Cycle 6 Day1, n=1, 0: number analyzed (Participants) | 1 | 0
  Magnesium, Cycle 6 Day1, n=1, 0 | 0.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. |

29. Secondary Outcome: Change From Baseline in Weight During Extension Phase
Description: Weight was measured at indicated time-points. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 6 | 2
Kilograms
  Cycle 2 Day 1, n=6, 2 | -1.6 (1.74) | -4.6 (4.31)
  Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Cycle 3 Day 1, n=3, 1 | -0.3 (1.00) | -4.5 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 4 Day 1, n=3, 0 | -2.3 (0.85) |
  Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 5 Day 1, n=3, 0 | -3.3 (2.91) |
  Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Cycle 6 Day1, n=2, 0 | -0.4 (0.92) |

30. Secondary Outcome: Change From Baseline in SBP and DBP During Extension Phase
Description: Vital signs including SBP and DBP were measured at indicated time-points. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 6 | 2
Millimeters of mercury
  DBP, Cycle 2 Day 1, n=6, 2 | -0.2 (3.19) | -12.0 (12.73)
  DBP, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  DBP, Cycle 3 Day 1, n=3, 1 | 8.7 (9.81) | -9.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  DBP, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  DBP, Cycle 4 Day 1, n=3, 0 | -0.3 (3.06) |
  DBP, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  DBP, Cycle 5 Day 1, n=3, 0 | 12.3 (6.51) |
  DBP, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  DBP, Cycle 6 Day1, n=2, 0 | 6.5 (4.95) |
  SBP, Cycle 2 Day 1, n=6, 2 | -1.2 (12.89) | -2.5 (23.33)
  SBP, Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  SBP, Cycle 3 Day 1, n=3, 1 | 6.7 (10.97) | -6.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  SBP, Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  SBP, Cycle 4 Day 1, n=3, 0 | -2.3 (7.57) |
  SBP, Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  SBP, Cycle 5 Day 1, n=3, 0 | 5.7 (10.02) |
  SBP, Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  SBP, Cycle 6 Day1, n=2, 0 | 13.0 (1.41) |

31. Secondary Outcome: Change From Baseline in Pulse Rate During Extension Phase
Description: Vital sign including pulse rate was measured at indicated time-points. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 6 | 2
Beats per minute
  Cycle 2 Day 1, n=6, 2 | 17.2 (10.15) | 9.0 (5.66)
  Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Cycle 3 Day 1, n=3, 1 | 23.0 (20.78) | 4.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 4 Day 1, n=3, 0 | 15.3 (8.08) |
  Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 5 Day 1, n=3, 0 | 9.3 (11.55) |
  Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Cycle 6 Day1, n=2, 0 | 16.5 (9.19) |

32. Secondary Outcome: Change From Baseline in Temperature During Extension Phase
Description: Vital sign including temperature was measured at indicated time-points. Baseline is defined as the most recent measurement prior to the first administration of study drug in extension phase. Change from Baseline was calculated as post dose value minus Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1 (each cycle was of 28 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Participants With Normal Hepatic Function | Participants With Impaired Hepatic Function
Number analyzed (Participants) | 6 | 2
Degrees Celsius
  Cycle 2 Day 1, n=6, 2 | -0.3 (0.77) | 0.1 (0.07)
  Cycle 3 Day 1, n=3, 1: number analyzed (Participants) | 3 | 1
  Cycle 3 Day 1, n=3, 1 | -0.1 (0.26) | 0.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Cycle 4 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 4 Day 1, n=3, 0 | -0.0 (0.38) |
  Cycle 5 Day 1, n=3, 0: number analyzed (Participants) | 3 | 0
  Cycle 5 Day 1, n=3, 0 | -0.1 (0.21) |
  Cycle 6 Day1, n=2, 0: number analyzed (Participants) | 2 | 0
  Cycle 6 Day1, n=2, 0 | -0.3 (0.21) |

ADVERSE EVENTS:
Time Frame: All cause mortality, non-SAEs and SAEs were reported from start of study treatment and up to Day 8 in PK Phase and up to 28 months in Extension Phase.
Description: All cause mortality, non-SAEs and SAEs were reported for Safety Population consisting of all participants who received atleast 1 dose of the investigational drug, niraparib. The results are presented based on final analysis up to 28 months.
Groups:
- Participants With Normal Hepatic Function-PK Phase; Participants With Normal Hepatic Function-Extension Phase: All participants received a single dose of 300 milligrams (mg) (3X100 mg capsules) niraparib administered on Day 1 of PK phase. Upon entering extension phase, participants with screening actual body weight >= 77 kilograms (kg) and current platelet count of >=150,000 cells per microliter (c/μL) at C1D1 continued to receive niraparib 300 mg/day (3X100 mg) once daily (QD) on Day 1 of every cycle until treatment discontinuation(each cycle of 28-days). Participants with screening actual body weight < 77 kg and/or current platelet count of <150,000 c/μL continued to receive niraparib 200 mg (2X100 mg capsules) QD on Day 1 of every cycle until treatment discontinuation (each cycle of 28 days).
- Participants With Impaired Hepatic Function-PK Phase; Participants With Impaired Hepatic Function-Extension Phase: All participants received a single dose of 300 mg (3X100 mg capsules) niraparib administered on Day 1 of PK phase. Upon entering extension phase, participants received niraparib 200 mg (2X100 mg capsules) QD on Day 1 of every cycle until treatment discontinuation (each cycle of 28 days).
Arm/Group | Participants With Normal Hepatic Function-PK Phase | Participants With Impaired Hepatic Function-PK Phase | Participants With Normal Hepatic Function-Extension Phase | Participants With Impaired Hepatic Function-Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 2/8 | 4/7
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/8 | 3/8 | 2/7
Other Adverse Events (participants affected / at risk) | 5/9 | 3/8 | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Normal Hepatic Function-PK Phase (N=9) | Participants With Impaired Hepatic Function-PK Phase (N=8) | Participants With Normal Hepatic Function-Extension Phase (N=8) | Participants With Impaired Hepatic Function-Extension Phase (N=7)
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Normal Hepatic Function-PK Phase (N=9) | Participants With Impaired Hepatic Function-PK Phase (N=8) | Participants With Normal Hepatic Function-Extension Phase (N=8) | Participants With Impaired Hepatic Function-Extension Phase (N=7)
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 2
Amylase increased (Investigations) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT03359850/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT03359850/SAP_001.pdf